CLINICAL TRIAL: NCT05728983
Title: Insufficient Sleep and Dietary Choices: An Ecologically Valid Examination of the Decision Foundations of Eating Behaviors When Sleep Restricted
Brief Title: Sleep and Food-based Decision Making
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Appalachian State University (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SES 2018001
Record Dates: First submitted 2023-01-23; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Participants randomly assigned to the treatment group arm experience both a well-rested and sleep-restricted week during the study
  Interventions: Other: Sleep levels
- Control group (Placebo Comparator): Participants randomly assigned to the treatment group arm experience two well-rested weeks during the study (and they still have an ad lib sleep week in between the two well-rested weeks)
  Interventions: Other: Sleep levels

INTERVENTIONS:
Other: Sleep levels — Sleep levels are what the experimenter prescribes to participants in the study.

SUMMARY:
This study administers two prescribed sleep levels, each lasting one week, that participants will complete in their at-home environment. One week is a well-rested (8-9 hrs/night attempted sleep) and another is a sleep-restricted (5-6 hrs/night attempted sleep) condition. In between these two conditions is an ad lib sleep week. At the end of each treatment week, the participants come to a laboratory session to go through a series of decision making tasks. Participants also track dietary intake through the 3-week protocol using the ASA24 website.

This study was fully preregistered on the open science framework (OSF) has has registration DOI at https://doi.org/10.17605/OSF.IO/NSPRK

DETAILED DESCRIPTION:
THE PRELIMINARY SCREENING SURVEY:

This short demographic, sleep, and mood survey is administered at least twice a year by the investigator (Dickinson) on random subsets of students at his institution. This database survey had been ongoing for several years and has been approved under separate human subjects approval process, and has been used by the investigator (Dickinson) to recruit for a variety of "sleep and decision" research studies over the years.

This short survey provides sufficient information for the investigators to screen out individuals who self-report a sleep disorder, who are not within the 18-40 year old target age range for this study, who are at significant risk of major depressive or anxiety disorder (assessed using validated short-instruments). Viable participants who meet the inclusion criterion (usually, only about 2/3 of those who complete the survey) are randomly assigned to either the control condition or a particular ordering of the treatment condition (SR-WR or WR-SR), ex ante. Afterwards, these individuals are invited to participate in the experiment via email. (note, participants are NOT allowed to opt into a condition or treatment ordering to which they were not randomly assigned)

THE SLEEP PROTOCOL:

The basic sleep protocol will involve recruitment of a total of 130 participants. Participants are randomly assigned to the control condition (N=30) or the treatment condition (n=100). The investigators anticipate some attrition such that n>130 will be enrolled in the study to ultimately obtain n=130 participants who will have successfully completed the entire protocol.

Both conditions involve 3-weeks of at-home prescribed sleep levels for the participants. For the Control participants, week 1 prescribes 8-9 hours of attempted sleep per night for the 7 nights of that week (refer to this as a well-rested [WR] week). Week 3 for Control participants will be another prescribed WR week.

Treatment participants will be prescribed a WR week in week 1 or week 3 and a sleep-restricted (SR) week (5-6 hrs/night attempted sleep) then in week 3 or week 1. That is, treatment participants will be administered the treatment conditions either in SR-WR or in WR-SR order (counterbalanced across participants). For all participants (control and treatment), week 2 is an ad lib sleep week to wash out the treatment effects of week 1 before commencing the week 3 prescribed sleep level.

All participants will complete basic sleep diary records for the entire 3 weeks and will wear a validated sleep-tracking actigraphy device for the duration of the period. Objectively measured actigraphy sleep data will be scored using validated protocols.

The idea of the 3-week sleep protocol is to obtain within-participants measures of decision-making that will be assessed at the end of weeks 1 and 3 (the treatment weeks) with the participant in an experimentally manipulated state of well-restedness or chronic partial sleep restriction (similar to recommended WR levels and levels of SR common in many adult populations).

ADDITIONAL STUDY ELEMENTS In addition to decision making that will be assessed at the end of weeks 1 and 3 of the protocol (i.e., after each experimentally prescribed sleep week), participants will also complete daily food recalls of their dietary intake over the course of the 3-week protocol, as well as a short form of the International Physical Activity Questionnaire (IPAQ) and validated measures of cognitive and sleep function at the end of each week of the protocol. The IPAQ, as well as cognitive and sleep function assessments, will be administered online prior to the in-lab decision session at the end of each week (all three weeks). The daily food recalls will be completed online using the Automated Self-Administered 24-hour dietary assessment tool (ASA24).

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age

Exclusion Criteria:

* at risk of major depressive or anxiety disorder (from validated screener), self-reported or suspected sleep disorder, extreme diurnal preference type (from validated screener)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Food-Image based go no-go task: | 3 weeks
  This task is validated in the literature and available in Inquisit programmed form. It assesses inhibitory control in food related image selection (go) or non-selection (no-go) as compared to non-food related images
Food-image based Approach Avoidance task | 3 weeks
  This is a validated task available in Inquisit programmed form and it assess automatic processing to compare one's tendency to approach (pull image towards oneself on computer screen) or avoid (push image away from oneself on computer screen) images reflecting healthier versus less healthy foods
Food Choice Task | 3 weeks
  This task gives participants a short time span (e.g., 10 seconds) to select a set of food images to place in one's onscreen cart. Images includes healthier and unhealthy items.
Food preference (ratings) task | 3 weeks
  This just asks individual to report on a 0-100 scale how much they like various foods based on a displayed image of each (with higher numbers meaning the participant likes the item more)
Delay-discounting monetary choice task | 3 weeks
  This validated task asks one's preference of monetary amounts received today versus larger amounts received at some future point (e.g., 7 days, or 85 days later). Actual choices are paid out for a randomly selected subset of participants on a randomly selected trial (different trials vary the size of the monetary difference and the number of delays for the delayed reward).
Food information based confirmation bias task | 3 weeks
  This task assesses one's tendency to consider arguments regarding the healthiness or tastiness of food as more or less strong based on whether that participants dominant food ideology favors the consideration of healthiness or tastiness of food. The investigators have pilot tested and published a paper on this task.
Snack/drink auction task | 3 weeks
  In this task, participants are given a snack and a beverage as part of a decision session and allowed to bid on how much they would pay (or need to be paid) to exchange their snack or drink for a different snack or drink. Various combinations of snack auctions and drink auctions are considered in order to compare willingness to pay for healthier or less healthy snacks or drinks)
Story retelling task | 3 weeks
  This validated task presents participants with a short story that they are asked to retell so that we can assess preservation of key story details.
Dietary intakes | 3 weeks
  These data are gathered from daily dietary intakes input by participants on the ASA24 dietary recall website, which allows for separation of outcomes by various macronutrients.

SECONDARY OUTCOMES:
Psychomotor vigilance task | 3 weeks
  This validated task assesses reaction time
Karolinska sleepiness scale | 3 weeks
  This validated task assess subjective sleepiness (in the moment). This is assess at Baseline and at the decision sessions that occur during the protocol.
Objective Sleep duration | 3 weeks
  These data are collected from research-grade actigraphy devices worn by the participant.

OTHER OUTCOMES:
BMI | 1 day
  Body mass index is assessed by self reported height and weight. This is assessed only at Baseline at the beginning of the protocol.
Emotional Eating Scale | 1 day
  An 18-item validated instrument assessing one's emotional approach to food. This is assessed only at Baseline at the beginning of the protocol.
Current Future self scale | 3 weeks
  An image-based task asking how interconnected one see's his/her current self with his/herself in 10 years (the more interconnected, the more this has been tied to low future-discounting rates). This is assessed at baseline and at decision sessions during the protocol.
mood reports | 3 weeks
  Likert-scale self-report of how strongly one feels the following emotions: attentive, upset, alert, irritable, determined, nervous. This is assessed at baseline and at decision sessions during the protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Appalachian State University, Boone, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No identifiable data are shared with other researchers